CLINICAL TRIAL: NCT01195389
Title: A Randomized, Single-Blind, Placebo-Controlled Pilot Study to Evaluate the Safety and Efficacy of the Application of Magnetic Fields Using the Resonator for the Treatment of Alzheimer's Disease in Addition to Standard of Care
Brief Title: Safety and Efficacy Study of Magnetic Fields to Treat Alzheimer's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: pico-tesla Magnetic Therapies, LLC (Industry)
Responsible Party: Allen S. Braswell Jr. CEO, Pico-Tesla Magnetic Therapies, LLC
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USF #6178-P67865
Record Dates: First submitted 2010-09-01; First posted 2010-09-06 (Estimated); Last update posted 2011-07-08 (Estimated); Status verified 2011-06

CONDITIONS: Alzheimer's Dementia
Keywords: dementia; memory loss; cognitive decline
MeSH Terms: conditions — Alzheimer Disease; Dementia; Memory Disorders; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Resonator (Active Comparator): Treatment with active Resonator device using low level magnetic fields
  Interventions: Device: Resonator
- Placebo treatment (Placebo Comparator)
  Interventions: Device: Resonator

INTERVENTIONS:
Device: Resonator — Treatment group vs. Placebo group

SUMMARY:
The purpose of this study is to determine if low level magnetic fields can help to improve memory in patients diagnosed with Alzheimer's dementia.

DETAILED DESCRIPTION:
The purpose of this pilot study is to determine whether application of magnetic fields generated by the Resonator result in statistically significant improvements in cognitive functioning and memory in patients with a diagnosis of Alzheimer's dementia.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of Alzheimer's Disease appropriately documented by the patients physician and/or neurologist
* Documentation verifying that other generally recognized causes of dementia have been ruled out by prior physician evaluations
* Mild to Moderate Dementia, as evidenced by a score of not less than 12 nor greater than 26 on the Mini Mental Status Exam (MMSE).
* Subject is ambulatory.
* A Study Partner who can attend all study visits with the subject. Study Partner being defined as an adult who has at least 10 hours/week of contact with the subject, and can accompany the subject to all testing and treatment study visits.
* Stable "anti-dementia" medication regimen without significant side effects for at least 3 months, and on stable medication (unrelated to anti-dementia) without significant side effects for at least 1 month; willingness and ability to maintain the stable medication regimen throughout the course of the study.
* Willingness and ability to present to the testing center for all study evaluations
* Willingness and ability to present to the treatment center for all study treatments (exposure to the Resonator™)
* Willingness to maintain stable diet and activity regimen for the duration of the study.
* Willing and able to abstain from partaking in any non-essential (not physician ordered) existing or new treatments to improve cognition and mental functioning
* Willing and able to abstain from any medications that could affect cognition and mental functioning during the course of the study
* Male or female.
* Any ethnic background.
* Age 55 and older.

Exclusion Criteria:

* Change in anti-dementia medical regimen within 3 months prior to initiation of study.
* Confirmed diagnosis other non-Alzheimer's type of dementia
* Significant neurologic or psychiatric illness other than Alzheimer's disease
* Unstable cardiac disease, such as any history of cardiac arrhythmias (including atrial fibrillation, ventricular fibrillation, or irregular atrial-ventricular conduction time), or any incidences of congestive heart failure, or myocardial infarction, within the last six months.
* Previous surgical interventions involving prosthetics or implants comprised of ferrous metals, or pacemakers, vagus nerve stimulators, or other functional electrical stimulators such as those commonly used for pain.
* Reported consumption of more than 14 alcoholic drinks per week.
* Uncontrolled hypertension.
* Uncontrolled atrial fibrillation or other uncontrolled arrhythmias, e.g. tachycardia, bradycardia.
* Uncontrolled seizure disorder.
* History of seizures or usage of anti-seizure medications that, in the opinion of the investigator, participation in this trial would represent a risk to the subject.
* Uncontrolled, unstable, or untreated medical conditions which may significantly impact the subject's health or ability to complete the entire study, in the opinion of the investigator.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-10 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale-Cog (ADAS-cog) | end of treatment at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Smith, MD, Principal Investigator — University South Florida Health Byrd Alzheimer's Institute
Locations (1):
- USF Health Byrd Alzheimer's Institute, Tampa, Florida, United States